CLINICAL TRIAL: NCT07292922
Title: Digital-supported Orofacial Myofunctional Therapy in Subjects With Obstructive Sleep Apnoea: A Pilot Randomised Control Trial
Brief Title: Digital-supported Orofacial Myofunctional Therapy in Subjects With Obstructive Sleep Apnoea: A Pilot Randomized Control Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Agnes LAI Yuen Kwan, Associate Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 25-461
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Orofacial Myofunctional Therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control group (No Intervention): The control (waitlist) group will not receive any intervention within the study period
- The Intervention group (Active Comparator): The intervention group will participate in a 3-month digital-support Myofunctional Therapy program. This innovative program is designed to ensure proper exercise performance, enhance adherence, and provide real-time feedback to patients.
  Interventions: Behavioral: Digital-supported Orofacial Myofunctional Therapy

INTERVENTIONS:
Behavioral: Digital-supported Orofacial Myofunctional Therapy — The intervention include: (1) Five 30-minute d-MFT sessions; (2) two follow-up phone calls; and (3) facial and tongue exercise app for home practice.
  Arms: The Intervention group

SUMMARY:
This pilot study explores the feasibility, acceptability, and preliminary effectiveness of Digital-supported Orofacial Myofunctional Therapy (d-MFT), an innovative program combining facial recognition technology with evidence-based orofacial exercises for individuals with mild to moderate obstructive sleep apnoea (OSA). The d-MFT program aims to strengthen oropharyngeal muscles, improve airway function, and reduce OSA severity.

We expect that participants receiving 3-month d-MFT (n=30) will demonstrate greater improvements in OSA severity, sleep-related symptoms, and quality of life compared to those in the waitlist control group (n=30).

Feasibility and acceptability will be evaluated through outcome-based questionnaires and semi-structured interviews exploring participants' experiences, satisfaction, and perceived barriers to adherence.

DETAILED DESCRIPTION:
This pilot study investigates the feasibility, acceptability, and preliminary effectiveness of Digital-supported Orofacial Myofunctional Therapy (d-MFT), an innovative approach that integrates facial recognition technology with evidence-based orofacial exercises tailored for individuals with mild to moderate obstructive sleep apnoea (OSA). Rooted in Self-Determination Theory, the d-MFT program aims to strengthen oropharyngeal muscles, enhance airway function, and alleviate OSA severity. The intervention consists of five 30-minute sessions and two follow-up phone calls conducted over three months, all delivered through a dedicated mobile application that provides real-time feedback and tracks adherence.

The primary objectives of this research are twofold: first, to evaluate whether d-MFT effectively reduces OSA severity and associated symptoms, and second, to identify barriers and facilitators to its implementation in real-world settings. We hypothesize that participants who receive the d-MFT intervention will show greater improvements in OSA severity, sleep-related symptoms, and overall quality of life compared to those in the control group.

This randomized controlled trial will recruit 60 participants, divided into two groups of 30 each, all diagnosed with mild to moderate OSA (apnoea-hypopnea index [AHI] of 5-30 events per hour). Individuals with severe comorbidities or a history of OSA-related surgery will be excluded. The intervention group will engage with the d-MFT app daily for three months, while the control group will continue their usual care before transitioning to the intervention after the assessment.

Outcomes will be measured at baseline and after three months. Objective assessments will include polysomnography to evaluate the apnoea-hypopnea index, oxygen desaturation index, and snoring severity. Subjective evaluations will be conducted using standardized questionnaires such as the Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, and Functional Outcomes of Sleep Questionnaire, providing insights into daytime sleepiness, sleep quality, and quality of life. Additionally, oropharyngeal muscle function will be assessed through tongue pressure measurements. Adherence to the d-MFT program will be monitored using electronic logs within the app.

Feasibility and acceptability will be assessed through semi-structured interviews that explore participants' experiences, levels of satisfaction, and perceived barriers to adherence. For quantitative data analysis, linear mixed-effects models will be utilized to account for repeated measurements and potential confounders, while qualitative data will be analyzed through thematic content analysis.

This study represents a promising non-invasive alternative that addresses existing treatment challenges by employing technology-enhanced therapy aimed at improving both adherence and clinical outcomes. Ultimately, the findings from this pilot study have the potential to significantly advance the management of obstructive sleep apnoea through broader implementation of d-MFT.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above
* Diagnosed with mild to moderate Obstructive Sleep Apnoea, defined as: Apnoea-Hypopnea Index of 5-30 events per hour
* Indications for Continuous Positive Airway Pressure or oral appliance treatment, but unable to tolerate or decline these treatments
* Body Mass Index less than 30 kg/m2

Exclusion Criteria:

* Presence of obstructive nasal disease or significant nasal obstruction
* Unstable mental health issues
* History of stroke
* Unstable chronic respiratory, cardiac, neurological conditions
* Inability to provide informed consent
* Prior oral, pharyngeal, or maxillofacial surgical therapy for sleep apnoea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Programme satisfaction | month 3
  Outcome-based questions on satification on the program
Change in oxygen saturation | Baseline and month 3
  Measured by sleep test

SECONDARY OUTCOMES:
Change in respiratory Indices | Baseline, month 3
  Measured by sleep test
Change in snoring | Baseline, month 3
  Measured by sleep test
Change in sleep quality | Baseline, month 3
  Measured by Insomnia Severity Scale, a 7-item questionnaire that assesses the severity of insomnia symptoms. Scores ranged from 0 to 28, with cutoffs for no clinically significant insomnia (0-7), subthreshold insomnia (8-14), moderate clinical insomnia (15-21), and severe clinical insomnia (22-28).
Change in daily function | Baseline, month 3
  Measured by Functional Outcomes of Sleep Questionnaire (FOSQ-10). A self-reported questionnaire designed to access the impact of excessive sleepiness on multiple daily activities. It consists of 10 items that evaluate various dimensions of sleep-related functional outcomes. Each item is rated on a 4 to 5-point Likert scale, with higher scores indicating less difficulty and better functional status. The total score is calculated by averaging the responses and converting them to a scale ranging from 5 to 20, with lower scores suggesting that sleep disturbances significantly impair daily functioning.
Change in oropharyngeal muscle function | Baseline, month 3
  Measured by Tongue Pressure assessment, which is an objective assessment of oropharyngeal muscle function, indicating the strength of the tongue during contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — Hong Kong Metropolitan University

IPD SHARING:
Plan to Share IPD: Undecided
It has not been mentioned during the IRB application.